CLINICAL TRIAL: NCT02949453
Title: ACCeptation and Qualitative Evaluation of Phone-delivered Intervention To Prevent Suicide Reattempt
Brief Title: ACCeptation and Qualitative Evaluation of Phone-delivered Intervention
Acronym: ACCEPT-S
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hôpital le Vinatier (Other)
Collaborators: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2016-A00919-42
Record Dates: First submitted 2016-10-24; First posted 2016-10-31 (Estimated); Last update posted 2019-04-08 (Actual); Status verified 2018-04

CONDITIONS: Suicide
Keywords: suicide; prevention
MeSH Terms: conditions — Suicide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients after suicidal episode (Experimental): Patients receiving a telephone-delivered intervention after deliberate self-harm (DSH)
  Interventions: Behavioral: Semi-directed interview performed by a social sciences researcher

INTERVENTIONS:
Behavioral: Semi-directed interview performed by a social sciences researcher — Two semi-directed interviews performed by social sciences researcher:
  * first interview performed 6 weeks after the suicide attempt, in an suicide prevention unit, duration 1 to 1.5 hour
  * second interview performed 3 month after the suicide attempt, in a suicide prevention unit, duration 1 to 1.5 hour

SUMMARY:
Background: Previous suicide attempt is known to be a strong risk factor for repetition and repetition is common within the first year after an episode of deliberate self-harm (DSH). There has been growing interest in brief interventions for this population that are focused on maintaining long-term contact and/or offering re-engagement with services when needed. Despite telephone-delivered interventions have shown promising results in suicide reattempt prevention, subjective impact of such brief contact interventions and effectiveness mechanisms have never been evaluated.

DETAILED DESCRIPTION:
Semi-structured in-depth interviews with 20 patients previously receiving a telephone-delivered intervention from our team. Six weeks and 3 months after a DSH, people included in telephone-delivered process will be interviewed by a social science researcher. Qualitative analysis using thematic analysis will be independently performed by two researchers.

ELIGIBILITY:
Inclusion Criteria:

* Deliberate self-harm in the previous week,
* 18 years old and older,
* outpatient care orientation after discharge from emergency department

Exclusion Criteria:

* Difficulties in french language,
* mental retardation

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2017-03-03 (Actual); Primary Completion 2019-04-04 (Actual); Study Completion 2019-04-04 (Actual)

PRIMARY OUTCOMES:
Acceptation of a telephone-delivered intervention after deliberate self-harm(DSH) | change from baseline after the telephone intervention
  analyze the acceptability for suicidal patients in the reiteration of the suicide prevention procedure performed by telephone Callback

SECONDARY OUTCOMES:
Impact of telephone-delivered intervention after a deliberate self-harm (DSH) | 2 years
  through the evaluation of this device Callback, we will identify its impact on pipelines and post-crisis experiences

CONTACTS AND LOCATIONS:
Overall Officials: TERRA JEAN-LOUIS, PUPH, Principal Investigator — Centre Hospitalier le Vinatier
Locations (1):
- Hopital Vinatier, Bron, France

IPD SHARING:
Plan to Share IPD: No